CLINICAL TRIAL: NCT07320950
Title: Neuroprotective Effect of Neurotropin on Chronic Oxaliplatin-induced Neurotoxicity in Stage II and Stage III Colorectal Cancer Patients: a Randomized, Double-blind, Placebo-controlled, Parallel Grouping Multi-center Clinical Trial
Brief Title: Neuroprotective Effect of Neurotropin on Chronic OXA-induced Neurotoxicity in Stage II and Stage III CRC Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gong Chen, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B2020-061-01
Record Dates: First submitted 2022-01-04; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: Adverse event; Oxaliplatin; Neurotoxicity; Neurotropin; Management
MeSH Terms: conditions — Colorectal Neoplasms; Neurotoxicity Syndromes | interventions — neurotropin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Neurotropin 4 tablets/day (Experimental): All the patients in this group received neurotropin 4 tablets a day ( 2 tablets once , twice a day, p.o.) ,given for 21 days (day 1-21) while the patient receiving the Oxaliplatin chemotherapy regimen from day1 to day 21 each cycle, totally for 8 cycles.
  Interventions: Drug: Neurotropin
- Neurotropin 8 tablets/day (Experimental): All the patients in this group received neurotropin 8 tablets a day ( 4 tablets once , twice a day, p.o.) ,given for 21 days (day 1-21) while the patient receiving the Oxaliplatin chemotherapy regimen from day1 to day 21 each cycle, totally for 8 cycles.
  Interventions: Drug: Neurotropin
- Placebo (Placebo Comparator): All the patients in this group received placebo 8 tablets a day ( 4 tablets once , twice a day, p.o.) ,given for 21 days (day 1-21) while the patient receiving the Oxaliplatin chemotherapy regimen from day1 to day 21 each cycle, totally for 8 cycles.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Neurotropin — Participants would be assess the safety and evaluate the neurotoxicity after the last cycle of whole chemotherapy regimen.
  Arms: Neurotropin 4 tablets/day; Neurotropin 8 tablets/day
Other: Placebo — placebo
  Arms: Placebo

SUMMARY:
Oxaliplatin is effective in adjuvant and first-line colorectal cancer chemotherapy. Oxaliplatin-induced severe chronic neurotoxicity is the main dose-limiting adverse event. No standard treatment for oxaliplatin-induced chronic toxicity has been defined. Neurotropin has been identified as a strategy for reducing the peripheral neurotoxicity in the published studies. Our aim is to define the best intake dose and evaluate the safety of neurotropin for peripheral neurotoxicity of oxaliplatin by conducting a placebo-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old
* Stage II or III colorectal cancer patients confirmed by pathological diagnosis, and recovered from surgery within 8 weeks
* should receive adjuvant chemotherapy especially XELOX regimen after assessment by physicians and specialists
* Agreed and assigned the consent, and was able to receive the baseline assessment
* Could be inpatient or outpatient participants

Exclusion Criteria:

* Peripheral neuropathy patients, e.g. diabetes neuropathy
* Alcoholic related patients
* Central neuropathy patients
* Patients who were unable to assess the effectivity and safety
* Neurotropin allergy
* History of medications that are contraindicated to neurotropin <28 days before the trial begins
* Have already received neurotropin tablets more than 4 tablets or 3.6 units <4 weeks before the trials begins
* Unable to visit the hospital regularly
* Has been ruled out by investigators
* Brain tumor or metastasis
* Brain injury, stroke and brain hemorrhage symptoms occurred during 6 months after sign the consent
* History of epilepsy, convulsion
* Severe respiratory, cardiovascular, renal, hepatic or hematologic system(except cancer) disease
* Depression and other psychologic conditions which investigators recognized as high risk for the enrollment
* Chronic pain
* Received other medication from other clinical trials within 28 days
* Prepare for pregnancy, pregnant, or lactated women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
The incidence of peripheral neurotoxicity among groups | At the end of chemotherapy (up to 8 cycles, each cycle is 21 days)
  Oxaliplatin specific neurotoxicity grade classification and assessment. Incidence of Grade 3 or higher peripheral neuropathy at the end of adjuvant chemotherapy

SECONDARY OUTCOMES:
The completion rate of oxaliplatin based chemotherapy | At the end of chemotherapy (up to 8 cycles, each cycle is 21 days)
  Calculate the exact cycles that the participants completed
Fine motor functions assessment | From completion of adjuvant chemotherapy, assessed at 2 years.
  Questionaire to assess whether the patient could complete the fine movement such as writing and zip up
Time from total recovery from neurotoxicity after the chemotherapy | From completion of chemotherapy, up to 3 years.
  The time (in months) from the first documented complete resolution of chemotherapy-induced peripheral neuropathy. Participants without recurrence will be censored at the date of last follow-up within the 3-year study period.
Disease-Free Survival (DFS) Rate at 3 Years | From randomization up to 3 years
  The proportion of participants who are alive and free of disease (i.e., have not experienced disease recurrence or a new primary cancer) at 3 years from the date of randomization (or start of treatment).
Overall Survival (OS) Rate at 3 Years | From randomization up to 3 years
  OS is defined as the time from the date of randomization to the date of death from any cause. Participants who are still alive at the time of analysis will be censored at the last known alive date.

CONTACTS AND LOCATIONS:
Overall Officials: Gong Chen, Prof, Principal Investigator — Sun Yat-sen University; Zhi-zhong Pan, Prof, Study Chair — Sun Yat-sen University; De-Sen Wan, Prof, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China